CLINICAL TRIAL: NCT06973486
Title: The Effects of Social, Emotional and Attitudinal Dynamics on Spinal Anesthesia Outcomes in Cesarean Delivery
Brief Title: Causes of Spinal Failure in Cesarean Section
Status: Not yet recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Yilmaz Guler, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: SF-2019
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Causes of Spinal Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: psychometric scales — Perceived Stress Scale (PSS) Pain Tolerance Scale (PRS) Surgical Anxiety Scale

SUMMARY:
The main purpose of this research is to determine the causes of spinal anesthesia failures during cesarean section due to social, emotional and attitude factors towards surgery and to use this information to improve anesthesia practice.

ELIGIBILITY:
Inclusion Criteria:

* spinal anesthesia for term pregnancy and cesarean section
* age ≥ 18
* knowing the gestational week when participating in the study
* answering all research questions
* using the internet and social media tools

Exclusion Criteria:

* mental and physical disability
* diagnosis and treatment for psychiatric disorders
* clinically significant physical health problemı

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women over 18 years of age receiving spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
spinal anesthesia success rate | 20 minute
  Causes of spinal anesthesia failure during cesarean section related to social, emotional and attitude factors towards surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714